CLINICAL TRIAL: NCT06105996
Title: ADIE-FS - Aligning Dimensions of Interoceptive Experience in Patients With Functional Seizures
Acronym: ADIE-FS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 155563; 322599 (Other: IRAS); 23/NS/0075 (Other: REC)
Record Dates: First submitted 2023-10-09; First posted 2023-10-30 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Psychogenic Nonepileptic Seizures; Dissociative Seizures; Psychogenic Pseudoseizure; Functional Neurological Disorder; Non Epileptic Seizure
Keywords: interoception; functional seizures; functional neurological disorder
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Conversion Disorder; Seizures

STUDY DESIGN:
Intervention Model Description: Participants in the study will be randomised to the intervention group (interoceptive training) or the treatment as usual group.
Who Masked: Outcomes Assessor
Masking Description: Participants will be assessed at the end of the study by members of the research team who have been blinded to whether the participant was randomised to the intervention group of the study, or the treatment as usual group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interoceptive training (Experimental): Participants will undergo 6 sessions of cardiac interoceptive training.
  Interventions: Behavioral: Interoceptive training
- Treatment as usual arm (No Intervention): Participants will undergo treatment as usual.

INTERVENTIONS:
Behavioral: Interoceptive training — There will be 6 interoceptive training sessions carried out over two months. Each training session will comprise two blocks, between which participants will undergo a self-paced, light physical activity that aims to enhance heartbeat perception and lasts 2 to 3 minutes. During the pre- and post-exercise block, each participant will complete cardiac interoceptive tasks, and for each trial, note their confidence in their answer on a visual analogue scale and then be given accurate feedback about their objective heartbeat perception accuracy and the accuracy of their subjective confidence rating, relative to their objective accuracy.
  Arms: Interoceptive training

SUMMARY:
Functional seizures are common and harmful. They look like epileptic seizures but are not caused by the excess electrical discharges in the brain that arise in epilepsy. Our understanding of the mechanisms that give rise to functional seizures is limited, and for this reason the development of novel treatments for functional seizures is also limited. Recent research by our and other groups has shown that interoception may play an important role in the development of functional seizures. Interoception refers to the process by which the nervous system senses, interprets and integrates information from inside the body. Research has shown that altered interoception is linked to functional seizures. We have shown that patients with functional seizures have a reduced ability to accurately identify signals from within their bodies, such as their heartbeats. The worse their ability, the greater their seizure severity and higher their levels of other unwanted symptoms. In separate research other groups have shown that interoceptive training, that is actively training an individual to better recognise signals from their body, can reduce levels of anxiety and the levels of unwanted symptoms. In this study we therefore plan to explore the feasibility of interoceptive training in patients with functional seizures.

DETAILED DESCRIPTION:
Functional seizures are common and harmful. They look like epileptic seizures but are not caused by the excess electrical discharges in the brain that arise in epilepsy. Recent research by our and other groups has shown that interoception may play an important role in the development of functional seizures. Interoception refers to the process by which the nervous system senses, interprets and integrates information from inside the body. Research using heartbeat recognition tests has shown that persons with functional seizures have a reduced ability to accurately read out signals originating from within their body, and that this corresponds with seizure frequency and other symptomatology. Separate research has shown that actively training an individual interoceptively using cardiac interoceptive tasks can reduce anxiety levels and somatic symptoms.

The primary objective of this study is to demonstrate the feasibility of an interoceptive therapy program to reduce functional seizure severity and/or duration for patients. The secondary objective is to ascertain if the interoceptive therapy program leads to an improvement in interoceptive measurements, health-related quality of life, exercise, psychosocial functioning, psychiatric symptoms, psychological distress, and somatic symptom benefit for patients.

This is an open label, feasibility and pilot study. There will be two arms, an intervention arm and a treatment as usual arm. We aim to recruit 10 participants in each arm (n=20 in total).

Participants with functional seizures will be recruited from UCLH (University College London Hospitals) neurology services. At an initial face-to-face meeting participants will sign the consent form and complete further questionnaires, in addition to those they have already completed at home. Participants will then be randomised to one of two groups, an intervention group and treatment as usual group. Participants in both groups will complete two cardiac interoceptive tasks at baseline. A schedule for the six interoceptive training sessions will then be agreed for those participants in the intervention group, and completed within two months. During each training session the participant will complete the cardiac interoceptive tasks with active feedback, before and after a 2 to 3 minute period of self-directed exercise whose purpose is to elevate the heartbeat. The purpose of the exercise is ultimately to increase cardiovascular arousal and accompanying sensations such that it is easier for them to perceive their heartbeat in the interoceptive tasks.

After the final training session, participants in both groups will complete the same set of questionnaires, and have one further face-to-face meeting, where they will complete the cardiac interoceptive tasks again. Participants in both groups will also be followed up at 3 months and repeat both the questionnaires and interoceptive testing.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Capacity to complete informed consent to take part in study
* Possible, or probable or clinically established or documented functional seizure as per International League Against Epilepsy (ILAE) criteria

Exclusion Criteria:

* Age below 18 years
* Past moderate to severe head injury as defined by Mayo criteria
* Moderate to severe cognitive impairment
* Co-existing or past neurological disorder causing sensorimotor symptoms
* Co-existing major psychiatric disorder with active psychosis
* Moderate to severe musculo-skeletal disease (e.g., osteoarthritis or rheumatoid arthritis) causing functional impairment (e.g., in gait or basic activities of daily living)
* Current substance or alcohol dependence
* A recent cardiovascular event (last 12 months) or undiagnosed chest pain
* BMI (body mass index > 40kg/m2)
* Taking cardiac ionotropic drugs
* Uncontrolled hypertension
* Pregnancy
* Uncontrolled asthma or COPD (chronic obstructive pulmonary disease)
* Are having cognitive behavioural therapy (CBT) specifically for functional seizures, or are due to have CBT specifically for functional seizures within the period of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with functional seizures who are eligible for our pilot study who agree to be enrolled in intervention arm of ADIE-FS. | 24 months
  Feasibility measure
Proportion of participants who complete the ADIE-FS programme of treatment. | 24 months
  Feasibility measure
Proportion of participants with a 3-item Client Satisfaction Questionnaire (CSQ-3) score ≥ 9 for the ADIE-FS intervention (range of scores is 8 to 32 where higher scores indicate increased satisfaction). | 24 months
  Feasibility measure
Proportion of participants taking part in intervention with a mean score on the Treatment Expectancy Questionnaire (TEQ) ≥ 50% for the ADIE-FS intervention (higher scores indicate greater expectancy that the intervention will be useful). | 24 months
  Feasibility measure

SECONDARY OUTCOMES:
Cardiac interoceptive accuracy scores | 24 months
  Changes in cardiac interoceptive accuracy scores from baseline to end of study will be calculated in both groups using behavioural tests. Higher scores will indicate greater objective interoceptive accuracy.
Cardiac interoceptive sensibility scores | 24 months
  Changes in cardiac interoceptive sensibility scores from baseline to end of study will be calculated in both groups using the Porges body awareness questionnaire. Higher scores will indicate greater subjective perception of interoceptive accuracy.
Cardiac interoceptive awareness scores | 24 months
  Changes in cardiac interoceptive awareness scores from baseline to end of study will be calculated in both groups. Higher scores will indicate lesser discrepancy between subjective and objective interoceptive accuracy.
Seizure frequency and bothersomeness | 24 months
  Changes in seizure frequency and bothersomeness from baseline to the end of the study will be calculated in both groups using seizure diaries and a seizure severity scale. Higher scores will indicate greater seizure frequency and severity.
Levels of physical activity. | 24 months
  Changes in levels of physical activity from baseline to the end of the study will be calculated in both groups using the International Physical Activity Questionnaire. Higher scores will indicate greater levels of physical activity.
Levels of detachment dissociation. | 24 months
  Changes in levels of trait detachment dissociation from baseline to the end of the study will be calculated in both groups using the multiscale dissociation inventory. Higher scores indicate greater levels of dissociation.
Levels of compartmentalisation dissociation. | 24 months
  Changes in levels of trait compartmentalisation dissociation from baseline to the end of the study will be calculated in both groups using the somatoform dissociation questionnaire. Higher scores indicate greater levels of dissociation.
Levels of anxiety. | 24 months
  Changes in levels of trait anxiety from baseline to the end of the study will be calculated in both groups using the trait anxiety inventory. Higher scores indicate greater levels of anxiety.
Levels of somatic symptoms. | 24 months
  Changes in levels of somatic symptoms from baseline to the end of the study will be calculated in both groups using the patient health questionnaire-15. Higher scores indicate greater levels of somatic symptoms.
Quality of life metric. | 24 months
  Changes in quality of life from baseline to the end of the study will be calculated in both groups using the 12 item short form survey. Higher scores indicate poorer quality of life.
Functional impairment. | 24 months
  Changes in functional impairment from baseline to the end of the study will be calculated in both groups using the work and social adjustment scale. Higher scores indicate greater functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Mahinda Yogarajah, PHD, Principal Investigator — UCL/UCLH
Locations (1):
- Queen Square Institute of Neurology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koreki A, Garfkinel SN, Mula M, Agrawal N, Cope S, Eilon T, Gould Van Praag C, Critchley HD, Edwards M, Yogarajah M. Trait and state interoceptive abnormalities are associated with dissociation and seizure frequency in patients with functional seizures. Epilepsia. 2020 Jun;61(6):1156-1165. doi: 10.1111/epi.16532. Epub 2020 Jun 5. PMID 32501547
- [Result] Quadt L, Garfinkel SN, Mulcahy JS, Larsson DE, Silva M, Jones AM, Strauss C, Critchley HD. Interoceptive training to target anxiety in autistic adults (ADIE): A single-center, superiority randomized controlled trial. EClinicalMedicine. 2021 Aug 1;39:101042. doi: 10.1016/j.eclinm.2021.101042. eCollection 2021 Sep. PMID 34401684